CLINICAL TRIAL: NCT07091734
Title: Tirzepatide for Partial Lipodystrophy Treatment: A New Horizon in 2024
Acronym: TILT-2024
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elif Oral, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUM00251971
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Lipodystrophy, Partial
Keywords: Tirzepatide
MeSH Terms: conditions — Lipodystrophy, Partial, Acquired | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled, open label, delayed onset cross-over study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirzepatide then usual care (Group A) (Experimental): Participants will have a 12-week run-in period and then recheck of eligibility. Eligible participants randomized to this group will receive Tirzepatide according to the dose titration plan described in the FDA-approved Prescribing Information (starting with 2.5 mg/week and increasing the dose every 4 weeks by increments of 2.5 milligrams (mg) for 24 weeks (up to 15 mg over the course of 6 months). Phase 2 weeks 25-48: Discontinuation of Tirzepatide (patients may continue on protocol if commercial use of GLP-1 receptor agonist is begun during this phase). Participants will continue the regular diabetic and hypertriglyceridemia medications that were used during the run-in period for weeks 25-48.
  Interventions: Drug: Tirzepatide; Drug: Usual care medications
- Usual care treatment then Tirzepatide (Group B) (Experimental): Participants will have a 12-week run-in period and then recheck of eligibility. Eligible participants randomized to this group will continue participant's regular diabetic and hypertriglyceridemia medications that were used during the run-in period for 24 weeks. During weeks 25-48 (phase 2) participants will receive Tirzepatide according to the dose titration plan described in the FDA-approved Prescribing Information (starting with 2.5 mg/week and increasing the dose every 4 weeks by increments of 2.5 milligrams (mg) for 24 weeks.
  Interventions: Drug: Tirzepatide; Drug: Usual care medications

INTERVENTIONS:
Drug: Tirzepatide — Participants will receive study drug (Tirzepatide) according to the dose titration plan described in the FDA-approved Prescribing Information (starting with 2.5 mg/wk and increasing the dose every 4 weeks by increments of 2.5 mg.
  Additionally, participants will have visits (virtual or remote visits every four weeks) as well as various tests and evaluations during the trial.
  Other Names: Mounjaro
Drug: Usual care medications — Participant's will continue on participant's regular diabetic and hypertriglyceridemia medications that were used during the run-in period for 24 weeks. This will be either Phase 1 or Phase 2 based on randomization.
  Additionally, participants will have visits (virtual or remote visits every four weeks) as well as various tests and evaluations during the trial.

SUMMARY:
This study aims to see if the clinical use of Tirzepatide in patients with lipodystrophy (a rare disorder associated with abnormal loss of the body's fat tissue) may lead to improved diabetes mellitus control and lowering of participant's triglycerides through the reduction of caloric intake.

Study Hypothesis:

- The clinical use of Tirzepatide in patients with lipodystrophy may lead to favorable outcomes through the reduction of caloric intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥18 years old) with a diagnosis of familial partial lipodystrophy (per protocol)
* Hemoglobin A1c ≥ 7.0% at screening and after 12-week run-in period and
* Triglycerides ≥ 200 Milligrams Per Deciliter (mg/dL) at screening and after 12-week run-in period
* Stable body weight during the 3 months prior to screening visit (no gain or loss of >5% current body weight)
* Diet must have been stable for the prior 3 months (i.e., no major change in macronutrient composition, e.g. starting or stopping diets such as Atkins, paleo, vegetarianism, veganism)
* Patients must be willing and able to comply with clinic visits and study-related procedures (if patients cannot complete clinical outcomes assessments or unable to undergo magnetic resonance imaging (MRI), participants will not necessarily be excluded)

Exclusion Criteria:

* Diagnosis of generalized lipodystrophy or acquired lipodystrophy
* Having received treatment with a Glucagon-like peptide (GLP) -1 agonist or Tirzepatide within the past 6 months
* History of previous treatment with metreleptin within the past 3 months
* Pancreatitis within the past 3 months
* Patients with a medical history of bone morrow transplant, use of an immune check-point inhibitor, or central nervous system tumor involving the hypothalamus
* Treatment with of receiving over the counter or prescription medications for weight loss within 3 months prior to the screening visit
* Active treatment with oral glucocorticoids >7.5 milligram (mg) prednisone equivalents per day or plans to begin treatment with oral glucocorticoids >7.5 mg prednisone equivalents per day during the study period
* Treatment with oral estrogens, aromatase inhibitors, Luteinizing hormone-releasing hormone (LHRH) agonists or systemic testosterone begun within 6 months prior to the screening visit
* Any malignancy, e.g., lymphoma, within the past 1 year, prior to screening visit except for fully treated basal cell or squamous epithelial cell carcinomas of the skin or carcinoma in situ of the cervix or anus
* A personal or family history of medullary thyroid carcinoma (MTC) or in patients with multiple endocrine neoplasia Type 2 (MEN 2)
* History of heart failure hospitalization, myocardial infarction, stroke, clinically significant arrhythmia (e.g., ventricular tachycardia, or any arrhythmia requiring medication adjustment to control), transient ischemic attack, unstable angina, percutaneous or surgical revascularization procedure (coronary, carotid, or peripheral vascular), or intracardiac device placement (e.g., pacemaker) within 3 months before the screening visit
* Advanced heart failure (New York Heart Association Class 3 to 4) or severe and uncontrolled hypertension
* Current diagnosis of autoimmune Type 1 diabetes mellitus
* History of human immunodeficiency virus (HIV) positivity or HIV positive at screening (to exclude HIV associated lipodystrophy).
* Uncontrolled infection with hepatitis B or hepatitis C infection or known active tuberculosis by history at screening
* A patient that has a documented, positive reverse-transcriptase polymerase chain reaction (RT-PCR) or serology test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) may be enrolled provided the patient has recovered from Coronavirus disease (COVID-19) (all COVID-19-related symptoms and have no major clinical findings which can potentially affect the safety of the patient)
* Participation in any clinical research study evaluating an investigational product (IP) or therapy within 3 months and less than 5 half-lives of IP prior to the screening visit. Participation in clinical research studies that only involve procedures (e.g., muscle biopsies, glycemic clamps) or testing (eg, MRI) that will not interfere with the current study is permitted
* Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study
* Alcohol consumption >21 drinks per week for males or >14 drinks per week for females
* Pregnant or breastfeeding persons. Patients, if engaged in sexual relations with/and of childbearing potential, must agree to use a highly effective contraceptive method from the time of signing the informed consent form until at least 4 weeks after the last dose of study drug
* Sexually active adult men that are unwilling to use the following forms of medically acceptable birth control during the study drug treatment period and for 16 weeks after the last dose of study drug: vasectomy with medical assessment of surgical success OR consistent use of a condom. Sperm donation is prohibited during the study and for 16 weeks after the last dose of study drug
* Known serious hypersensitivity to Tirzepatide or any of the excipients in Mounjaro

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) from baseline in Group A (Tirzepatide-treated) versus Group B (control) at 24 weeks | Baseline, 24 weeks
  Height and weight will be collected to calculate BMI.
Change in Hemoglobin A1c from baseline in Group A (Tirzepatide-treated) versus Group B (control) at 24 weeks | Baseline, 24 weeks
  The A1c is a blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Oral, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication of data shall occur during the project, if appropriate, or at the end of the project, consistent with normal scientific practices. Research data that documents, supports, and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. Such research data will be redacted to prevent the disclosure of personal identifiers.
  The study data will be submitted to the Central Biorepository at the University of Michigan or the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository when appropriate. Transcriptomic datasets that can be shared will be deposited in Gene Expression Omnibus (GEO, National Center for Biotechnology Information). Clinical and phenotypic datasets will be associated with the ribonucleic acid (RNA) sequencing submission to GEO.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award. The study data will be stored in the repository for at least 5 years.
Access Criteria: In accordance with federal regulation and institutional policies, data and associated documentation will be available to users only under a data-sharing agreement that provides for (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. A standard data use agreement has been developed by the University and will be used. In addition, all data-sharing arrangements must comply with institutional policies, which are subject to change. The study team have included the plan to share data with other investigators in our consent forms